CLINICAL TRIAL: NCT04799834
Title: Study of the Genetic Factors That Influence the Susceptibility to and Severity of COVID-19
Brief Title: Genotype and Susceptibility to COVID-19
Acronym: ORIGIN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: ORIGIN
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Covid19
Keywords: COVID-19; Genotype
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CASES: Subjects who have had a severe form of COVID-19 and developed respiratory failure requiring oxygen supplementation or CPAP mechanical ventilation or intubation
  Interventions: Other: Questionnaire administration,blood sampling and genetic analyses.
- CONTROLS 1: Subjects, comparable in age, sex and risk factors (such as concomitant diseases) with the CASES, who contracted the virus but either did not fall ill or had mild symptoms
  Interventions: Other: Questionnaire administration,blood sampling and genetic analyses.
- CONTROLS 2: Subjects, comparable in age, sex and risk factors (such as concomitant pathologies) with the CASES, who did not contract the virus
  Interventions: Other: Questionnaire administration,blood sampling and genetic analyses.

INTERVENTIONS:
Other: Questionnaire administration,blood sampling and genetic analyses. — Adults (≥18 years) living in Bergamo and in all the towns of its territory shall be invited to voluntarily complete a questionnaire, with their personal data and information on SARS-CoV-2 clinical history (swab test and serologic test results, clinical symptoms, treatments, hospital care) and other previous conditions. Subjects considered fit for the genetic study will be asked to report to the Daccò Clinical Center for an interview, during which the data entered in the questionnaire will be reviewed and implemented, the informed consent for participation in the genetic investigations will be collected and blood sampling will be carried out.
  Genetic: Exome sequencing and genotyping of host genome of individuals infected with SARS-CoV-2 and showing severe disease (cases), or infected with SARS-CoV-2 and showing mild disease or remaining asymptomatic, and in individuals without evidence of infection with SARS-CoV-2 (negative sierology).

SUMMARY:
COVID-19 is a viral disease induced by infection with the novel SARS-CoV-2 coronavirus. Infection arises from the inhalation of viral particles spread by an infected individual. The main virus entry pathways are the nose and mouth mucous membranes, particularly rich in ACE2 receptors, that are used by the virus to enter cells and begin its replication.

Not all individuals who contract the virus fall ill, and most of those who do (about 70-80%) experience mild symptoms (fever, cough, headache, muscle aches, loss of taste and smell). If the immune system is unable to rapidly fight the virus back, the latter can attack the lungs, affeting oxygen absorption inside the alveoli and lead to pneumonia. This more severe form is observed in 20% of patients and can develop into even more serious complications requiring intensive care, with a high mortality rate. In severe cases (about 5%), the disease spreads to the entire body reaching the cardiovascular system and brain, with the risk of heart attacks, encephalitis and stroke, but it can also affect the liver, kidney and bowel.

Reasons why some subjects develop a highly severe disease while others have little or no symptoms at all still remain unclear. Many researchers are trying to find an answer by investigating the human genome, and the Mario Negri laboratories are also working in this direction.

The general hypothesis underlying this research project is that inter-individual genetic variations can explain the different responses to viral infection in a population, and that COVID-19 severity is, therefore, genetically determined in each infected subject.

ELIGIBILITY:
Inclusion Criteria:

- Age > 18 years

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) living in Bergamo and in all the towns of its territory
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Identification of the genetic determinants of COVID-19 severity. | Through study completion, an average of 10 months.
  Identification of variants in one or more candidate gene(s) responsible for the severe manifestation of COVID-19.
Identification of genetic factors affecting risk of SARS-Cov-2 infection. | Through study completion, an average of 10 months.

SECONDARY OUTCOMES:
Identification of polymorphic variants or mutations affecting treatment response in severe COVID-19 patients. | Through study completion, an average of 10 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro di Ricerche Cliniche per le Malattie Rare "Aldo e Cele Daccò", Ranica, BG, Italy